CLINICAL TRIAL: NCT01799278
Title: A Phase II Trial of the Aurora Kinase A Inhibitor MLN8237 in Patients With Metastatic Castrate Resistant and Neuroendocrine Prostate Cancer
Brief Title: A Phase II Trial of MLN8237 in Patients With Metastatic Castrate Resistant and Neuroendocrine Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1210013164
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Small Cell Prostate Cancer; Neuroendocrine Prostate Cancer; Prostate Adenocarcinoma Plus > 50% Immunohistochemical Staining for Neuroendocrine Markers
Keywords: Metastatic prostate carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): MLN8237 at 50 mg twice daily for 7 days repeated every 21 days. Therapy will continue until disease progression, unacceptable toxicity as a result of MLN8237, or withdrawal of patient consent.
  Interventions: Drug: MLN8237

INTERVENTIONS:
Drug: MLN8237 — MLN8237 will be administered orally. The study drug will be administered on an empty stomach with the patient remaining nothing by mouth (NPO), except for water and prescribed medications, for 2 hours before and 1 hour after each dose. Patients will be instructed to take each oral dose of MLN8237 with 8 ounces (1 cup, 240 mL) of water.
  Other Names: Alisertib

SUMMARY:
This study will evaluate the response rate of MLN8237 in patients with histologically confirmed or clinically suspected metastatic neuroendocrine prostate cancer (NEPC). MLN8237 is an orally administered Aurora kinase A inhibitor that has demonstrated broad antitumor activity in vitro and in vivo. In preclinical models, aurora kinase inhibition resulted in dramatic and preferential anti-tumor activity in NEPC with suppression of neuroendocrine marker expression.

DETAILED DESCRIPTION:
This is a multi-institutional single-arm, open-label Phase 2 trial evaluating MLN8237 in patients with histologically confirmed or clinically suspected metastatic neuroendocrine prostate cancer. Subjects will be treated with MLN8237 at 50 mg twice daily for 7 days repeated every 21 days. Individual dose reductions will be made on the basis of the AEs observed. Therapy will continue until disease progression, unacceptable toxicity as a result of MLN8237, or withdrawal of patient consent. Patients will be followed with history, physical, and blood tests at each visit to monitor for toxicity. Response and progression will be evaluated by CT/MRI scan and bone scan after every 3 cycles and determined using RECIST v1.1. PSA and serum chromogranin A and NSE will be followed every cycle. CTC counts by CellSearch will be performed at baseline, at 4-6 weeks, and upon progression. Patients will be followed for survival endpoints following completion of this study until death.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic prostate carcinoma and at least one of the following:

  * Histologic diagnosis of small cell or neuroendocrine prostate cancer
  * Histologic diagnosis of prostate adenocarcinoma plus > 50% immunohistochemical staining for neuroendocrine markers (chromogranin, synaptophysin or neuron specific enolase)
  * Development of liver metastases in the absence of PSA progression as defined by PCWG2
* Serum chromogranin A level >5 x upper limit of normal and/or serum neuron specific enolase (NSE) >2x upper limit of normal
* Measurable disease by RECIST 1.1 with PCWG2 modifications
* Patients with pure small cell neuroendocrine carcinoma on histology are not required to have received prior androgen deprivation therapy (ADT) or castrate levels of testosterone, but their testosterone state should be maintained for the duration of the study. Other patients are required to have surgical or ongoing chemical castration, with baseline testosterone level <50ng/dL.
* Patients capable of fathering children must agree to use an effective method of contraception for the duration of the trial and should continue use for 4 months after last dose of study drug
* Subjects must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration.
* ANC > 1500/mm³, platelets > 100,000/mm³, Hgb > 9 g/dL. Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days, however, erythrocyte growth factor is allowed as per published ASCO guidelines.
* Total bilirubin ≤ ULN, SGOT (AST) and SGPT (ALT)< 1.5 x ULN. AST and/or ALT may be up to 5X ULN if with known liver metastases provided bilirubin is normal.
* Adequate renal function as defined by serum creatinine ≤ 1.5 x ULN. If creatinine >1.5 x ULN, calculated or measured creatinine clearance must be ≥ 40 mL/minute (Cockcroft-Gault).
* ECOG performance status 0-2
* Estimated life expectancy > 3 months
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Radiation therapy to 25% of bone marrow within 2 weeks of first dose
* Residual > Grade 2 toxicity from prior treatment must have resolved with the exception of those explicitly described elsewhere in entry criteria
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen.
* Requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids or H2 antagonists are allowed (see section 5.5)
* Severe or uncontrolled systemic infection
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
* Currently active other malignancy excluding controlled non-melanoma skin cancer. Patients are considered NOT to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.
* Treatment with the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himisha Beltran, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (8):
- United States (8):
  - University of Chicago, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beltran H, Oromendia C, Danila DC, Montgomery B, Hoimes C, Szmulewitz RZ, Vaishampayan U, Armstrong AJ, Stein M, Pinski J, Mosquera JM, Sailer V, Bareja R, Romanel A, Gumpeni N, Sboner A, Dardenne E, Puca L, Prandi D, Rubin MA, Scher HI, Rickman DS, Demichelis F, Nanus DM, Ballman KV, Tagawa ST. A Phase II Trial of the Aurora Kinase A Inhibitor Alisertib for Patients with Castration-resistant and Neuroendocrine Prostate Cancer: Efficacy and Biomarkers. Clin Cancer Res. 2019 Jan 1;25(1):43-51. doi: 10.1158/1078-0432.CCR-18-1912. Epub 2018 Sep 19. PMID 30232224

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: MLN8237 at 50 mg twice daily for 7 days repeated every 21 days.
Period: Overall Study
Arm/Group | All Patients
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: This is a single-arm, open-label Phase 2 trial evaluating MLN8237 in patients with histologically confirmed or clinically suspected metastatic neuroendocrine prostate cancer. Subjects will be treated with MLN8237 at 50 mg twice daily for 7 days repeated every 21 days. Individual dose reductions will be made on the basis of the AEs observed. Therapy will continue until disease progression, unacceptable toxicity as a result of MLN8237, or withdrawal of patient consent
Arm/Group | All Patients
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 67 [45 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects are Male
  Participants
    Female | 0
    Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Response Rate, as Assessed by CT/MRI and Bone Scan, of Treatment With MLN8237 for Patients With Neuroendocrine Prostate Cancer
Description: Evaluated per RECIST 1.1 guidelines: Complete response (CR) is defined as complete disappearance of all measurable and evaluable lesions by physical examination or imaging studies and normalization of PSA with no appearance of new lesions for > 1 month. Partial response (PR) is defined as a 30% 56 or greater reduction in the sum longest unidimensional diameter of all measurable lesions. There may be no new lesions. Stable Disease (SD) is characterized by patients who do not meet the criteria of PR and who are without signs of progressive disease for at least 1 month. Disease Progression (DP) is defined as a greater than 20% increase in the sum longest unidimensional diameters of the indicator lesions or the appearance of new lesions. Bone scan progression (evaluable disease only) is defined by PCWG2 criteria. Per consensus guidelines in CRPC, to be considered measurable, lymph nodes need to be at least 2 cm in greatest dimension and 1.5 cm in short axis.
Time Frame: one year
Measure: Number; unit: participants
Groups:
- All Patients: MLN8237 at 50 mg twice daily for 7 days repeated every 21 days. Therapy will continue until disease progression, unacceptable toxicity as a result of MLN8237, or withdrawal of patient consent. MLN8237: MLN8237 will be administered orally. The study drug will be administered on an empty stomach with the patient remaining nothing by mouth (NPO), except for water and prescribed medications, for 2 hours before and 1 hour after each dose. Patients will be instructed to take each oral dose of MLN8237 with 8 ounces (1 cup, 240 mL) of water.
Arm/Group | All Patients
Number analyzed (Participants) | 60
participants | 18

2. Secondary Outcome: Progression-free Survival in Response to Therapy
Description: Patients will be followed for survival endpoints following completion of this study until death.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ALL SUBJECTS: A single-arm, open-label Phase 2 trial evaluating MLN8237 in patients with histologically confirmed or clinically suspected metastatic neuroendocrine prostate cancer. Subjects will be treated with MLN8237 at 50 mg twice daily for 7 days repeated every 21 days.
Arm/Group | ALL SUBJECTS
Number analyzed (Participants) | 60
months
  Castration-Resistant Prostate Cancer | 2.2 [2.0 to 2.6]
  Neuroendocrine Prostate Cancer | 2.3 [2.0 to 2.6]
  Castration-Resistant ProstateCancer-Adenocarcinoma | 2.0 [2.0 to 2.6]

3. Secondary Outcome: Overall Survival in Response to Therapy
Description: Patients will be followed for survival endpoints following completion of this study until death
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 60
months | 9.5 [7.4 to 13.0]

4. Secondary Outcome: Prostate-Specific Antigen (PSA) Test Response Rate
Description: PSA to be followed every cycle to determine response.
Time Frame: 2 years
Population: Data were not collected for this outcome.
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Circulating Tumor Cell (CTC) Response
Description: CTC counts by CellSearch will be performed at baseline, at 4-6 weeks, and upon progression to determine response.
Time Frame: 2 years
Population: Data were not collected for this outcome.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs which are serious must be reported to WCMC from first dose of MLN8237 up to and including 30 days after administration of the last dose of MLN8237. When possible, signs and symptoms indicating a common underlying pathology should be noted as one comprehensive event.
Description: An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a product whether or not it is related to the medicinal product. For this protocol an abnormal laboratory value will not be assessed as an AE unless that value leads to discontinuation or delay in treatment, dose modification, therapeutic intervention, or is considered by the investigator to be a clinically significant change from baseline.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 48/60
Serious Adverse Events (participants affected / at risk) | 23/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=60)
Neutropenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 6
Pain (General disorders) | 1
Electrolyte abnormalities (Metabolism and nutrition disorders) | 4
Infection (urinary tract, skin) (Renal and urinary disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Rash (Immune system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=60)
Fatigue (General disorders) | 47
Anorexia (Gastrointestinal disorders) | 27
nausea (Gastrointestinal disorders) | 23
pain (General disorders) | 23
Dyspnea (Immune system disorders) | 16
Alopecia (Skin and subcutaneous tissue disorders) | 16
Depression (Psychiatric disorders) | 13
Urinary frequency (Renal and urinary disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Edema (Ear and labyrinth disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Hematuria (Renal and urinary disorders) | 10
Dizziness (Ear and labyrinth disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 8
Hot flashes (Vascular disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Fever (General disorders) | 7
Creatinine increased (Investigations) | 7
Peripheral sensory neuropathy (General disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-05-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT01799278/Prot_000.pdf